CLINICAL TRIAL: NCT05545722
Title: The Effect of Life Coaching With Diabetes on Glycemic Control, Strengthening Diabetes and Self-management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuğba Bilgehan (Other)
Responsible Party: Sponsor-Investigator, Tuğba Bilgehan, Research Assistant, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-20
Record Dates: First submitted 2022-05-22; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus; Nurse-Patient Relations; Nurse's Role
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- life coaching group with diabetes (Experimental): Individuals with diabetes in the intervention 1 group will be interviewed for 'life coaching with diabetes'. Coaching is a set of systems that make people think deeply and reveal their own awareness and potential. A coach is a person who deliberately applies all these systems with awareness. Life coaching sessions with diabetes are based on the philosophy of coaching. Sessions are continued with questions that will enable the individual to realize the deficiencies in diabetes self-management. It helps the person with diabetes to discover solutions.This training will last for 3 months, once in 10 days. A total of 9 interviews will be provided.
  Interventions: Behavioral: life coaching group with diabetes
- Standard diabetes education (Experimental): Standard diabetes education will be given to individuals with diabetes in this group. This training will last for 3 months, once in 10 days. A total of 9 interviews will be provided.
  Interventions: Behavioral: life coaching group with diabetes
- control group (No Intervention): only pre-test and post-test were applied to this group. The patients in this group are the patient group who received training from the diabetes nurse of the hospital.

INTERVENTIONS:
Behavioral: life coaching group with diabetes — Each patient was interviewed once a week. Coaching interviews were conducted one-on-one and in accordance with coaching principles.
  Arms: Standard diabetes education; life coaching group with diabetes

SUMMARY:
Diabetes Mellitus (DM) is an endocrine and metabolic disease that is characterized by hyperglycemia, develops microvascular and macrovascular complications, and requires chronic and continuous care. is a disease. According to IDF 2019 data, it is predicted that the number of diabetics in the world, which was 463 million in 2019, will reach 700 million in 2045 with an increase of 51%. The global prevalence of diabetes between the ages of 20-79 in 2019 is 9.3%, and it is estimated to increase to 10.2% in 2030 and 10.9% in 2045. Our country, on the other hand, has the highest prevalence with a rate of 11.1% among European countries. According to the IDF 2019 Diabetes Atlas data, 6.6 million people with diabetes live in our country as of 2019, and it is estimated that this rate will reach 10 million by 2045.

American Diabetes Association (American Diabetes Association) and American Association of Clinical Endocrinologists (American Association of Clinical Endocrinologists) to achieve the goals of treatment and care in individuals with diabetes; emphasizes the need for regulation of nutrition, regulation of physical activity, regulation of pharmacological treatment, diabetes education, continuous monitoring and health controls. Individuals with diabetes should receive diabetes self-management education and support when necessary. Diabetes self-management is defined as the process of facilitating the knowledge, skills and abilities necessary for the individual's self-care. Individuals with diabetes who are competent and skilled in self-management can improve their health outcomes. The American Diabetes Association (ADA) defines diabetes self-management education as a process that begins at the diagnosis stage and continues, based on an individual-centered approach and making joint decisions to facilitate the knowledge, skills and abilities necessary for the self-care of diabetes patients.

The purpose of diabetes self-management is for diabetics to develop new skills and behaviors that support self-management goals, and to form habits. The general goals of diabetes self-management education are to support individuals diagnosed with diabetes to make conscious decisions, solve problems, perform self-care behaviors, and improve their metabolic results, health status and quality of life. Diabetes patients need knowledge, skills and motivation to strengthen their diabetes by providing self-management. The nurse helps the patient to adapt to the disease and achieve the ability to perform self-care by counseling and training individuals. Coaching sessions are used to strengthen self-management and diabetes in diabetes. The coach is the person who provides the necessary motivation to maximize the strengths of the client, to ensure that the potentials are fully used through continuous education, to develop new skills and activities to be more effective, to be ready for new responsibilities and to manage himself. Life Coaching with Diabetes is based on the basic principles and principles of professional life coaching practices (ICF-International Coaching Federation), aiming at behavioral change in approaches related to diabetes lifestyle. Life coaching with diabetes is to give practical applications to people who have been diagnosed with diabetes in order to gain necessary changes in life through coaching.

2. Problem and Sub-Problems H0: Diabetes life coaching given to individuals with Type 2 Diabetes has no effect on glycemic control, diabetes strengthening and self-management.

H1: Diabetes life coaching given to individuals with Type 2 Diabetes has an effect on glycemic control, strengthening diabetes and self-management.

3. Aims and Expected Benefits of the Research This study was planned as a control group intervention study to determine the effect of diabetes coaching on glycemic control, diabetes strengthening and self-management in individuals with Type 2 Diabetes.

Expected benefits:

* Developing appropriate self-care activities (physical activity, medical nutrition, drug management, avoiding risky behaviors, etc.) by improving the self-management skills of the individual with diabetes,
* Individuals with diabetes become self-managed in their self-care practices,
* Ensuring metabolic control of the diabetic individual
* Developing decision-making and problem-solving skills of individuals with diabetes,
* Promoting diabetes coaching in the nursing profession and increasing its visibility and spreading diabetes coaching.

DETAILED DESCRIPTION:
Research Method In the study, data will be collected by means of the data collection form, the diabetes strengthening scale, the diabetes self-management scale in people with type 2 diabetes, and based on the researcher's experiences and literature.

1. Data collection form: It will be created by the researcher based on the literature. (such as age, gender, how many years have had diabetes).
2. Diabetes strengthening scale: It has 3 sub-dimensions: management of psychosocial aspects in diabetes, level of dissatisfaction and readiness for change, setting and achieving diabetes goals.
3. Diabetes self-management scale for people with type 2 diabetes: The scale developed by has 3 sub-dimensions: healthy lifestyle, blood sugar management, and use of health services. High scores on the scale indicate good self-management, and low scores indicate poor self-management.

ELIGIBILITY:
Inclusion Criteria:

* The patient;

  * Being between the ages of 18-65,
  * Being literate,
  * Having a smart phone and being able to use it actively,
  * Having been diagnosed with type 2 diabetes at least 1 year ago,
  * No chronic complications related to diabetes have developed,
  * HbA1c > 7,
  * Absence of any psychiatric or mental problems,
  * Having the cognitive competence to answer questions,
  * Willingness to participate in the research

Exclusion Criteria:

* • The patient's desire to leave the study,

  * Inability to reach the patient by phone
  * Having advanced retinopathy, nephropathy, neuropathy, foot wound,
  * Being pregnant,
  * Being diagnosed with cancer, having myocardial infarction in the last 3 months,
  * Having type 1 diabetes.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 102 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
diabetes self-management skill scale | 12 weeks
  Diabetes self-management scale in people with type 2 diabetes: The score that can be obtained from the scale is between 95-19. A high score from the scale indicates good self-management, and a low score indicates poor self-management.

SECONDARY OUTCOMES:
Diabetes strengthening scale | 12 weeks
  Diabetes strengthening scale: The maximum score that can be obtained from the scale is 140, and the minimum score is 28. High scores in scale scoring indicate high levels of reinforcement; low scores indicate low levels of empowerment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tuğba Bilgehan, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bilgehan T, Vardar Inkaya B. The effect of a holistic nurse coaching intervention on glycemic control, diabetes self-management, and empowerment: a randomized controlled trial. BMC Nurs. 2025 Jun 2;24(1):627. doi: 10.1186/s12912-025-03252-0. PMID 40457333